CLINICAL TRIAL: NCT02388022
Title: A Retrospective Study Using CALIBER® TLIF Expandable Spacer in the Treatment of DDD: 2 Year Follow-up.
Status: Completed | Type: Observational
Sponsor: Globus Medical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: RGC13-005-PL_A
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2015-03

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- degenerative disc disease: Patients who have had a transforaminal lumbar interbody fusion at 1-2 contiguous levels with the CALIBER® expandable spacer and have completed at least 2 year follow-up.
  Interventions: Device: Degenerative Disc Disease

INTERVENTIONS:
Device: Degenerative Disc Disease — lumbar interbody with posterior screw and rod instrumentation
  Other Names: CALIBER

SUMMARY:
The purpose of the study is to gather clinical and radiographic outcome data from patients who have undergone treatment with an expandable interbody spacer.

DETAILED DESCRIPTION:
This is a multi center retrospective study with 200 patients. Sites will screen their patient records for patients who have had a TLIF utilizing the CALIBER® expandable interbody spacer in conjunction with the REVOLVE® or REVERE® posterior stabilization systems and subsequent follow-up visits.

The study aims to collect both pre-operative and post-operative data at the 6, 12 and 24 month time points according to existing standard of care and the surgeon's custom and practice.

ELIGIBILITY:
Inclusion Criteria:

* Objective evidence of degenerative disc disease at 1 or 2 level(s) between L2 and S1 resulting from degeneration of disc confirmed by history and radiographic studies.
* At least 18 years of age and maximum 80 years of age

Exclusion Criteria:

* • Presence of systemic or localized infection at the site of surgery

  * More than 2 levels to be instrumented
  * Previous fusion attempt at the involved level(s)
  * Spondylolisthesis unable to be reduced to Grade 1
  * Previous documentation of osteopenia, osteoporosis, or osteomalacia to a degree that spinal instrumentation would be contraindicated
  * Diagnosis of a condition or on postoperative medication(s), which may interfere with bony/soft tissue healing
  * Presence of a disease entity or condition which totally precludes possibility of bony fusion (e.g. metastatic cancer, HIV, long term use of steroids, etc.)
  * History of substance abuse (drugs or alcohol)
  * Mentally incompetent or prisoner

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both male and female between the ages of 18 and 80 with objective evidence of degenerative disc disease between L2 and S1 at 1-2 contiguous levels.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
radiographic evaluation | Pre-Op to 2 years post-operative
  Standing anterior-posterior, lateral, flexion and extension images

SECONDARY OUTCOMES:
Clinical outcomes | pre-op to 2 years post-operative
  Visual Analog Scale, Oswestry Disability Index, Neurological Exam

CONTACTS AND LOCATIONS:
Overall Officials: Choll Kim, MD, Principal Investigator — Spine Institute of San Diego

IPD SHARING:
Plan to Share IPD: Yes
Once data collection is complete and analyzed, we will submit to journals for publication